CLINICAL TRIAL: NCT00485082
Title: Disclosure of a Cystic Fibrosis Diagnosis to a Dating Partner
Brief Title: Disclosing a Cystic Fibrosis Diagnosis to a Dating Partner
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999907162; 07-HG-N162
Record Dates: First submitted 2007-06-09; First posted 2007-06-12 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-08-25

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Disclosure; Dating Partner; Phone Interview
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
This study will examine the experience of disclosing a cystic fibrosis (CF) diagnosis to a dating partner. CF has implications for potential life partners (issues of fertility, decreased life span and an increasing need for medical management with age) that may make disclosure particularly sensitive. An understanding of the disclosure process may provide insight into ways health care practitioners can support their patients during this process.

People between 21 and 35 years of age with CF who have been in at least one dating relationship may be eligible for this study.

Participants are interviewed by telephone about their experiences living with cystic fibrosis and telling dating partners about their diagnosis. The interview includes questions about:

* Past experiences disclosing their CF diagnosis to a dating partner
* What information was disclosed versus what was not disclosed
* Why certain information was disclosed or not disclosed
* Positive and negative implications of the disclosure or non-disclosure

The interview lasts about 60 minutes and is tape-recorded for later review and analysis.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is an autosomal recessive chronic medical condition. As medical treatment is improving more persons with CF are living into adulthood and are entering into serious dating relationships. A diagnosis of CF has medical implications of concern to potential life partners including infertility, decreased life span and an increasing need for medical management with age. In addition, there is a small but non negligible possibility of future children inheriting the condition. These implications may make this type of disclosure a particularly important event in one's life and may affect one's disclosure decisions. Little research has been done on the process of disclosure in this population, and research specifically on disclosure to dating partners is lacking.

This study seeks to gain insight into the experience of disclosing a CF diagnosis to a dating partner through semi-structured in-depth phone interviews with approximately 30 persons who have CF and who vary in gender, age, ethnicity, and severity of their condition. The interviews will explore general experiences of disclosure to dating partners, will focus on selective disclosure of certain information to certain recipients, and will explore the implications of the disclosure or non-disclosure experiences. The qualitative interviews will be transcribed and subjected to thematic analysis, which will identify common themes across interviews. An understanding of the disclosure process experienced by persons with cystic fibrosis may provide insight into ways health care practitioners can support their patients during this process.

ELIGIBILITY:
* INCLUSION CRITERIA:

Self-reported to have been diagnosed with cystic fibrosis.

Self-reported to be in or have been in at least one dating relationship

English speaking.

EXCLUSION CRITERIA:

Younger than 21 years of age; Older than 35 years of age.

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50
Dates: Start 2007-06-05; Primary Completion 2008-03-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Holt R, Court P, Vedhara K, Nott KH, Holmes J, Snow MH. The role of disclosure in coping with HIV infection. AIDS Care. 1998 Feb;10(1):49-60. doi: 10.1080/09540129850124578. PMID 9536201
- [Background] Kalichman SC, DiMarco M, Austin J, Luke W, DiFonzo K. Stress, social support, and HIV-status disclosure to family and friends among HIV-positive men and women. J Behav Med. 2003 Aug;26(4):315-32. doi: 10.1023/a:1024252926930. PMID 12921006
- [Background] Joachim G, Acorn S. Life with a rare chronic disease: the scleroderma experience. J Adv Nurs. 2003 Jun;42(6):598-606. doi: 10.1046/j.1365-2648.2003.02663.x. PMID 12787233